CLINICAL TRIAL: NCT04812392
Title: The Impact of 3 Days of Reduced Physical Activity on Endothelial Function and Glycemic Control in Active Older Adults
Brief Title: Physical Inactivity Impacts on Blood Vessel Health and Glucose Levels in an Aging Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leryn Reynolds (Other)
Responsible Party: Sponsor-Investigator, Leryn Reynolds, Assistant Professor, Old Dominion University
Organization: Old Dominion University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ERP-2021-12576
Record Dates: First submitted 2021-03-16; First posted 2021-03-23 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Aging; Cardiovascular Diseases; Glucose Intolerance
Keywords: diabetes; physical inactivity; vascular function
MeSH Terms: conditions — Cardiovascular Diseases; Glucose Intolerance; Diabetes Mellitus; Sedentary Behavior | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Acute Physical Inactivity (Experimental): Subjects will undergo 3 days of reduced physical activity.
  Interventions: Device: Continuous Glucose Monitoring System

INTERVENTIONS:
Device: Continuous Glucose Monitoring System — Subjects will wear a continuous glucose monitoring system for 3 days during the 3 day reduced physical activity phase.

SUMMARY:
Physical inactivity is known to increase post meal blood sugar levels in young, active populations. However, how quickly this may occur in active, older adults is not clear. Further, the relationship between blood vessel health and blood sugar disturbances which occur to acute physical inactivity is not clear. It is unknown if impairments in blood vessel function precede increases in blood sugar levels that occurs with inactivity in an aging population. This study aims to determine if short term reductions in physical activity impair blood vessel health and blood glucose control to a greater extent in an aging population compared to a young population. The investigators hypothesize that 3 days of reduced physical activity will result in impaired blood vessel function and glycemic control in an aged population.

DETAILED DESCRIPTION:
Subjects will undergo testing in 2 study phases separated by at least 2 weeks: 1) active phase: subjects will have post meal glucose levels measured across 3 days of participating in their normal exercise routines. Blood vessel health will also be measured via flow mediated dilation at the end of the 3 day monitoring period. 2) physically inactive phase: subjects will stop participating in exercise for 3 days while post meal glucose levels are measured. Blood vessel health will also be assessed on days 1, 3 of removal of exercise. The subject will need to come into the lab on these days of inactivity to have blood vessel health measured.

The study procedures are described below.

Continuous Glucose Monitoring The investigators would like to gain more information about how blood sugar levels change over the course of a day in a free living setting. To do this the investigators will use a continuous glucose monitoring system (CGMS). This system is what individuals with diabetes frequently use to monitor their glucose levels over the course of the day. Subjects will be asked to wear the CGMS for 3 consecutive, full days on 2 different occasions. This includes 3 days during their normal regular physical activity, then for 3 days following during the no exercise protocol. The CGMS is worn on the stomach, and it is a tiny glucose sensor which is inserted just under the skin. This device measures and records blood glucose values throughout the day. In addition, subjects will be asked to make at least four finger stick blood glucose readings taken with a standard glucose meter at different times each day and record these numbers on a log sheet. During the continuous glucose monitoring, subjects will need to consume the same type and quantity of foods at the same time each day (i.e. whatever the subjects consumes on day 1 of baseline testing, they need to eat that exact same food, volume of food and at the same time on days 1-3 of the study). Meals and snacks consumed are also entered into a paper-based diary.

Blood Vessel Health Measurement (Flow Mediated Dilation: FMD) Subjects will be asked to perform their normal exercise routines 12-16 hours prior to blood vessel health being measured in the active phase as well as prior to the first blood vessel health measurement in the inactive phase to control for the acute effects of exercise on blood vessel health. Blood vessel health will be measured at the end of the active phase in both groups of subjects. Further blood vessel health will be measured following 1, 3 days of being inactive in both groups of subjects. Blood flow to the leg will be measured by applying blood pressure cuffs around the ankle. Pre flow mediated dilation diameter and velocity are recorded for 3 minutes prior to a blood pressure cuff being inflated for 5 minutes. Following cuff deflation, a 2-minute diameter and velocity recording is collected.

ELIGIBILITY:
Inclusion Criteria:

1. 55 years and older, 18-40 years old
2. Healthy, physically active, performing at least 90 min/week of physical activity
3. Free of physical limitations that may interfere with alterations in daily physical activity levels

Exclusion Criteria:

1. Physician diagnosed metabolic disease, HIV, hepatitis, or tuberculosis.
2. Body weight change of greater than 5% within the previous 2 months
3. Smoking within the previous 2 months.
4. Taking medications that alter blood glucose levels

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
Change in glycemic control during a reduced physical activity state | The change of blood glucose values from pre-inactivity and following 3 days of inactivity
  The change in blood glucose levels measured following consumption of a meal will be assessed before inactivity and following 3 days of inactivity.

CONTACTS AND LOCATIONS:
Overall Officials: Leryn Reynolds, Ph.D., Principal Investigator — Old Dominion University
Locations (1):
- Old Dominion University, Norfolk, Virginia, United States

IPD SHARING:
Plan to Share IPD: No